CLINICAL TRIAL: NCT02611401
Title: The Efficacy of a Mindfulness Based Intervention for Depressive Symptoms in Patients With Multiple Sclerosis and Their Caregivers. A Randomized Controlled Clinical Trial.
Brief Title: Efficacy of MBI for Depressive Symptoms in Patients With MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Principal Investigator, luca ostacoli, Dr., University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Turin
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis; Depression
Keywords: multiple sclerosis; depression; mindfulness
MeSH Terms: conditions — Multiple Sclerosis; Depression | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindulness Based Intervention (Experimental): intervention with group-based Mindfulness Based Intervention
  Interventions: Behavioral: Mindfulness
- Active Control (Active Comparator): intervention with group-based Psychoeducation and Relaxation
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness — The MBI is based on MBSR protocol but in order to maximize the clinical utility in people with MS suffering from depressive symptoms, we will tailor mindfulness intervention on the needs of this specific population. We will apply a modified MBSR protocol integrated with techniques from Sensorimotor Psychotherapy.
  The MBI comprises an 8-week group program. Participants will took part in a 3 hour single weekly sessions, and there will be also an additional all-day session of 7 hours. Each session will cover specific exercises and topics within the context of mindfulness practice and training. Participants will be required to carry out daily 45-min homework assignments, which consist on mindfulness exercises and mindfulness applications in everyday life.
  Arms: Mindulness Based Intervention
Behavioral: Psychoeducation — The control group is designed to control for the nonspecific elements of the MBI treatment. It will be based on a psycho-educational framework and will include some relaxation techniques. In each session is discussed a MS-related topic. Relaxation and gentle stretching exercises will be proposed at the end of each session. Homework and the material (photocopies, slides, etc.) discussed in group sessions is left to each participant to encourage participants to practice exercises between sessions.
  This intervention will follow the same structure and weekly format of the MBI intervention. The only difference will be the absence of an all-day session.
  Arms: Active Control

SUMMARY:
Multiple Sclerosis has a great impact on psychological functioning of patients and can be associated with various psychological disorders and symptoms. The most prevalent one is depression, which ranges from 15% to 47%. Mindfulness Based Intervention (MBI) is a relatively brief and cost-effective program that has been studied in patients with several diseases.

Aims. To evaluate the efficacy of a group-based MBI on depressive symptoms, QoL and on correlated symptoms of MS patients and their caregivers.

Methods. The study design is a randomized controlled clinical trial. The subjects of the study are 88 patients with MS and depressive symptoms that will be pre-screened from among a catchment group of about 500 patients using the Beck Depression Inventory-II (BDI). The 88 patients will subsequently be randomized into two groups (44 in the experimental group and 44 in the active control group). The psychological assessment, independent and blind to treatment, will be performed with the same timing and tools: at baseline (T0), after treatment (T1), and 6 months after the end of the group intervention (T2). The assessment will encompass the administration of the clinical interview and other self-report questionnaires.

The experimental group will undergo a 8 weekly sessions of 3 hours each (plus an all day session) with group based MBI. The MBI is an Mindfulness Based Stress Reduction protocol integrated with body centered techniques from Sensorimotor Psychotherapy, in order to better tailor it on the needs of people with MS suffering from depressive symptoms. The active control group is designed to control for the non-specific elements of the MBI treatment and will follow the same structure as the MBI. It will be based on a psycho-educational framework and will include relaxation techniques.

Primary outcome measures in patients will be: 1) the proportion of participants at T1 and T2 that does not have a BDI-II score greater than 13; 2) the proportion of patients no longer meeting the diagnostic criteria for mood disorders as assesses by the SCID; 3) the improvement of FAMS scores for the six primary aspects of QoL.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) can be associated with various psychological disorders and symptoms. Depression is present in about 15-47% of MS patients, and it is estimated to be three times greater than the general population.

Anxiety and depression are closely associated, both independently and in interaction, with fatigue. Mohr et al. (2003) have shown that improvements of depressive symptoms are closely associated with a decrease in the severity of fatigue. These symptoms represents the most disabling symptoms that have heavy psychosocial consequences for patients, for example affecting relationships, leisure activities and employment. Given also the young age at which MS occurs it is important that these symptoms be adequately recognized and treated to prevent their chronicity.

A recent study on psychological treatment of depressive symptoms in patients with medical disorders stated that treating comorbid depression should be one of the priorities in medical care settings. Feinstein (2011) highlighted that treatments for depression in public health care services may also be adjusted according to the availability of resources and access to them. Thereby it is essential to establish brief and cost-effective interventions to reduce depression symptoms and the psychological burden and to improve the Quality of Life (QoL) of these patients.

Mindfulness-based interventions have been proven effective in improving depressive symptoms and in enhancing QoL in many different chronic conditions and recently also in MS patients.

Mindfulness could be defined as a nonjudgmental awareness and acceptance of one's moment-to-moment experience. As described by Bishop et al. (2004), mindfulness consist of two main component: the self- regulation of attention and a particular orientation toward the experience. Self-regulation of attention concern the nonjudgmental observation and awareness of physical sensations, affective states and thoughts as they arise. Orientation to experience refers to the attitude of acceptance and curiosity toward one's experience. Mindfulness has an effect on the distressing tendencies to escape from or to over-engage with one's disturbing feelings and thoughts.

Several studies have highlighted the effects of mindfulness on psychological health: ithas been associated with higher levels of QoL, life satisfaction, self-esteem, empathy, self-compassion,sense of autonomy and competence among both clinical and non-clinical populations. In addition, thesestudies have shown a negative correlation between mindfulness and negative affect and psychopathologicalsymptoms, such as depressive symptoms, rumination, anger, difficulties in emotion regulation, and social anxiety.

These studies also showed the efficacy of MBI in improving anxiety and depression symptoms related with physical illnesses like cancer, chronic fatigue syndrome, fibromyalgia, chronic pain, arthritis, diabetes, heart disease, stroke, and traumatic brain injury.

Several studies of neuroimaging and on biological markers have also pointed out the effects of mindfulness on a neurobiological level, showing its effects on the regulation of emotional responses through the inhibition of amygdala by a proper functioning of the prefrontal cortex and in an altered cortisol and immune patterns consistent with less stress and mood disturbance, and decreased blood pressure.

In recent years, there has been a widespread of mindfulness-based approaches, generically called Mindfulness Based Intervention (MBI), that are based upon MBSR but also incorporate techniques derived from clinical psychology and psychotherapy, which mainly focus on emotion regulation, on the development of somatic resources, on self-compassion (directed both towards themselves and towards others, i.e. loving kindness and compassion meditation, and that have a greater focus than MBSR on mind-body integration and on interpersonal relationships.

MBI are considered as an effective and cost-effective treatment addressing the difficulties derived from the serious psycho-social impact of highly disabling chronic diseases, such as MS, by changing a range of emotional and evaluative dimensions that underlie general aspects of well-being. MBI can be therefore useful in counteract the suffering caused by the symptoms, the fatigue, the depressive and anxiety symptomatology and the distress in dealing with the disability. A key objective of the MBI interventions is the improvement of QoL.

Moreover, some studies reported that stress may be one factor that influences the risk of MS exacerbation. This highlights even more the importance of developing interventions aimed at reducing stress in patients with MS. The study of Grossman et al. (2010), to our knowledge the only study that evaluates the efficacy of a group MBI in MS by comparing it with the usual care, showed that a cost-effective and relatively brief group intervention may improve a broad range of parameters of well-being of patients with MS.

This study has some limitations that our research project aims to overcome, such as the lack of a control group to assess the specificity of MBI, and the lack of objective measures of emotional measures and psychopathological symptoms.

In our project, we propose to include an active control intervention (psycho-education plus relaxation) in addition to usual care, and to assess the psychological functioning of MS patients with a semi-structured clinical interview (SCID) in addition to the self-report measures.

Moreover, we aim to evaluate the efficacy of the MBI in MS patients who have depressive symptoms, measured as having a score greater than 13 at the Beck Depression Inventory-II. The NICE guidelines (2009) indicate that psychological interventions such as mindfulness or psycho-education, combined with drug therapies or alternative to them depending on the case, resulted more effective both in terms of efficacy and in term of cost-effectiveness compared to drug therapy alone. Also as highlighted by Hofmann et al., (2010) MBI may be more effective in populations with mood disorders.

Furthermore, our project aims to involve patients' caregivers asking them to participate in the group to which the patient has been assigned. We expect that caregivers will benefit from the treatment received, due to the load of stress and difficulties related to the management of a chronic disabling diseases like MS. Furthermore, a recent study has shown that patients' depressive state influenced the deterioration of QoL and the depression of caregivers. In fact the MBI does not deal directly with the disease, but with the attitude of relating to the self, the others and to life. Finally, our project is based on MBSR protocol but in order to maximize the clinical utility in people suffering from MS and depression, we tailored mindfulness intervention on the needs of this specific population. We will apply a modified MBSR protocol integrated with body centered techniques from Sensorimotor Psychotherapy (SP; Ogden et al., 2006). SP was developed by Pat Ogden on the model of Ron Kurtz, a body psychotherapy built on mindfulness (Kurtz, 1990). Most of these points are already part of the MBSR model, but in this integration they are deepened more specifically to increase the clinical efficacy.

We aim to evaluate whether a group-based Mindfulness Based Intervention can reduce depressive symptoms and improve the QoL of patients, also reducing correlated symptoms, like anxiety, fatigue and perceived stress and modifying the perception of the disease and how to deal with interpersonal relationships. Primary aim: to evaluate the efficacy of MBI on depressive symptoms and QoL of MS patients, compared to an active control intervention and to a usual care group, and to assess whether these expected benefits can be maintained at the 6-month follow-up.

The secondary aim of the study is to assess whether after the Mindfulness Based Intervention there is an improvement in anxiety symptoms, in fatigue and in perceived stress; another secondary aim is to evaluate the efficacy of the intervention on the perception of the illness and whether participating in the MBI improve also the interpersonal relationship. Another secondary aim is to evaluate the efficacy of MBI on depression, QoL and related symptoms in caregivers.

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of MS (Mc Donald Criteria) evaluated by a neurologist at least six months prior the beginning of the study;
* relapsing-remitting and secondary progressive disease;
* age 18-65 years old;
* clinically inactive phase of the disease ;
* a score >13 on the Beck Depression Inventory-II (according to Goldman Consensus Group, 2005);
* an Expanded Disability Status Scale (EDSS) score of =6;
* fluent Italian speaker;
* legal capacity to consent to the treatment;
* willingness to abstain from or to suspend all concomitant psychological treatment;
* suspension of all psychotropic medications at least one month before the treatment or maintenance at baseline level throughout the study.

Exclusion Criteria:

* current severe Major Depressive Disorder;
* severe suicidality, including ideation, plan, and intent;
* current serious psychological and psychiatric disorders, including psychotic disorders, bipolar disorders, active substance abuse (as assessed by the SCID);
* presence of overt dementia;
* corticosteroid treatment during the previous 30 days;
* other serious medical disorders in addition to MS;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
depression score | 6 months follow-up
  the proportion of participants at T2 that do not have a BDI-II score greater than 13

SECONDARY OUTCOMES:
mood disorder | 6 months follow-up
  the proportion of patients no longer meeting the diagnostic criteria for mood disorders as assesses by the SCID at T2
QoL | 6 months follow-up
  the improvement of FAMS scores for the six primary aspects of QoL at T2

CONTACTS AND LOCATIONS:
Overall Officials: luca ostacoli, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Clinical and Biological Sciences Department, Orbassano, Turin, Italy

REFERENCES:
- [Derived] Carletto S, Tesio V, Borghi M, Francone D, Scavelli F, Bertino G, Malucchi S, Bertolotto A, Oliva F, Torta R, Ostacoli L. The Effectiveness of a Body-Affective Mindfulness Intervention for Multiple Sclerosis Patients with Depressive Symptoms: A Randomized Controlled Clinical Trial. Front Psychol. 2017 Nov 30;8:2083. doi: 10.3389/fpsyg.2017.02083. eCollection 2017. PMID 29250012
- [Derived] Carletto S, Borghi M, Francone D, Scavelli F, Bertino G, Cavallo M, Malucchi S, Bertolotto A, Oliva F, Ostacoli L. The efficacy of a Mindfulness Based Intervention for depressive symptoms in patients with Multiple Sclerosis and their caregivers: study protocol for a randomized controlled clinical trial. BMC Neurol. 2016 Jan 13;16:7. doi: 10.1186/s12883-016-0528-0. PMID 26757728